CLINICAL TRIAL: NCT01922856
Title: A Phase 2b Controlled Efficacy Study of Intradermally Delivered ETEC Fimbrial Tip Adhesin Vaccine Against Experimental Challenge With ETEC H10407 in Healthy Adult Volunteers
Brief Title: Challenge Study of an ETEC Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-12-24; NMRC.2013.0011 (Other: NMRC IRB); CIR 289 (Other: CIR)
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Enteritis; Escherichia Coli, Enterotoxigenic
MeSH Terms: conditions — Enteritis; Escherichia coli Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Challenge (Vaccinated) (Experimental): The vaccine will be administered via the ID route to alternating upper arms on days 0, 21, and 42.
  On the morning of challenge, subjects will drink 120 mL of bicarbonate buffer. Approximately 1 minute later, subjects will drink a solution of virulent H10407 bacteria suspended in the remaining 30 mL of bicarbonate buffer (2 x 10P7P cfu).
  Interventions: Biological: LTR192G with dscCfaE
- Challenge (Unvaccinated) (Experimental): On the morning of challenge, subjects will drink 120 mL of bicarbonate buffer. Approximately 1 minute later, subjects will drink a solution of virulent H10407 bacteria suspended in the remaining 30 mL of bicarbonate buffer (2 x 10P7P cfu).
  Interventions: Other: No Intervention

INTERVENTIONS:
Biological: LTR192G with dscCfaE — Recombinant fimbrial adhesin (dscCfaE) with Modified Escherichia coli (E coli) heat labile enterotoxin (LTR192G)
  Arms: Challenge (Vaccinated)
Other: No Intervention — Controls only receive challenge
  Arms: Challenge (Unvaccinated)

SUMMARY:
The purpose of the study is to determine the efficacy of a vaccine against enterotoxigenic E. coli (ETEC)-caused diarrhea.

DETAILED DESCRIPTION:
The purpose of the study is to establish preliminary efficacy of dscCfaE administered with LTR192G by intradermal (ID) immunization in prevention of disease caused by a challenge with a CFA/I expressing ETEC strain (H10407).

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 through 50 years (inclusive).
* General good health, without clinically significant medical history, physical examination findings or clinical laboratory abnormalities per clinical judgment of PI.
* Negative pregnancy test. Pregnancy at any time will result in not receiving any or additional investigational product. Females of childbearing potential must agree to use an efficacious hormonal or barrier method of birth control during the study. Abstinence is acceptable. Female subjects unable to bear children must have this documented (eg, tubal ligation or hysterectomy) or must have negative pregnancy tests.
* Willingness to participate in the study after all aspects of the protocol have been explained and written informed consent obtained.
* Completion of a training session and demonstrated comprehension of the protocol procedures, knowledge of ETEC-associated illness, and by passing a written examination (70% passing score).
* Availability for the study duration, including all planned follow-up visits.

Exclusion Criteria:

General

* Presence of a significant medical or psychiatric condition which in the opinion of the investigator precludes participation in the study. Some medical conditions which are adequately treated and stable would not preclude entry into the study. These conditions might include stable asthma controlled with inhalers or mild hypertension stably controlled with a single agent.
* Significant abnormalities in screening hematology, or serum chemistry as determined by PI or PI in consultation with the research monitor and sponsor.
* Presence in the serum of HIV antibody, HBsAg, or HCV antibody.
* Evidence of IgA deficiency (serum IgA < 7 mg/dL or below the limit of detection of assay).
* Evidence of current excessive alcohol consumption or drug dependence (a targeted drug screen may be used to evaluate at the clinician's discretion).
* Evidence of impaired immune function.
* Recent vaccination or receipt of an investigational product (within 30 days before vaccination).
* Any other criteria which, in the investigator's opinion, would compromise the ability of the subject to participate in the study, the safety of the study, or the results of the study

Research Related Exclusions Applicable to Vaccination and Challenge Participation

* History of microbiologically confirmed ETEC or cholera infection in last 3 years.
* Occupation involving handling of ETEC or Vibrio cholerae currently, or in the past 3 years.
* Symptoms consistent with Travelers' Diarrhea concurrent with travel to countries where ETEC infection is endemic (most of the developing world) within 3 years prior to dosing, OR planned travel to endemic countries during the length of the study.
* Vaccination for or ingestion of ETEC, cholera, or E coli heat labile toxin within 3 years prior to dosing.

Research Related Exclusions Not Applicable to Challenge-Only Participants

* Exclusionary skin history/findings that would confound assessment or prevent appropriate local monitoring of AEs, or possibly increase the risk of an AE.
* History of chronic skin disease (clinician judgment).- History of atopy such as active eczema.
* Acute skin infection/eruptions on the upper arms including fungal infections, severe acne, or active contact dermatitis.
* History of significant allergic reactions to any vaccines and allergies that may increase the risk of AEs (Well-controlled seasonal allergies responsive to antihistamine medication or intranasal steroids are not exclusionary per clinician determination).

Study-specific Exclusion Criteria

* Abnormal stool pattern (fewer than 3 per week or more than 3 per day).
* Regular use of laxatives, antacids, or other agents to lower stomach acidity.
* Use of any medication known to affect the immune function (eg, systemic corticosteroids and others) within 30 days preceding the first vaccination or planned use during the active study period.
* Known allergy to two of the following antibiotics: ciprofloxacin, trimethoprim-sulfamethoxazole, and penicillin.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2013-09-19 (Actual); Primary Completion 2016-02-06 (Actual); Study Completion 2016-07-14 (Actual)

PRIMARY OUTCOMES:
Number of adverse events associated with vaccine | Up to 1 year
Number of prevented diarrhea episodes | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar Talaat, MD, Principal Investigator — Johns Hopkins Center for Immunization Research
Locations (2):
- United States (2):
  - Johns Hopkins Center for Immunization Research, Baltimore, Maryland
  - Naval Medical Research Center, Silver Spring, Maryland